CLINICAL TRIAL: NCT00041379
Title: Phase I/II Study to Assess the Safety and Efficacy of Low Doses of Beta LT in Patients With Waldenstrom's Macroglobulinemia
Brief Title: Beta Alethine in Treating Patients With Waldenstrom's Macroglobulinemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LifeTime Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069494; LIFETIME-LTP-01-03
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2005-12

CONDITIONS: Lymphoma
Keywords: Waldenström macroglobulinemia
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia | interventions — alethine

INTERVENTIONS:
Drug: beta alethine

SUMMARY:
RATIONALE: Biological therapies such as beta alethine use different ways to stimulate the immune system and stop cancer cells from growing.

PURPOSE: Phase I/II trial to study the effectiveness of beta alethine in treating patients who have Waldenstrom's macroglobulinemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor effects of low-dose beta alethine in patients with Waldenstrom's macroglobulinemia.
* Determine the effects of this drug on anemia, performance status, and disease symptoms in these patients.
* Determine the effects of this drug on the immune system of these patients.
* Determine the safety of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive beta alethine subcutaneously on days 1, 15, 29, 43, 57, and 71. Courses repeat every 85 days in the absence of disease progression or unacceptable toxicity.

Patients are followed for 30 days.

PROJECTED ACCRUAL: A total of 13-37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of Waldenstrom's macroglobulinemia

  * Urine or serum protein electrophoresis showing a measurable monoclonal spike
  * Indolent disease not yet requiring therapy allowed
* Positive delayed-type hypersensitivity (DTH) response

  * Induration greater than 2 mm for at least 1 antigen
* No clinical signs or evidence of active brain involvement or leptomeningeal disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 50-100%

Life expectancy:

* At least 4 months

Hematopoietic:

* Neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 10 g/dL

Hepatic:

* Albumin at least 3.5 g/dL
* Bilirubin less than 2.0 mg/dL
* Transaminases no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No acute changes on EKG
* No uncontrolled angina
* No heart failure
* No arrhythmia

Other:

* Adequate nutritional intake as evidenced by total protein at least 60 g/L
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No concurrent gastrointestinal bleed
* No active bacterial infections such as abscess or with fistulae
* HIV negative
* No other concurrent non-malignant disease that would preclude study
* No history of alcoholism, drug addiction, or psychotic disorders that would preclude follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* More than 4 weeks since prior immunotherapy
* More than 4 weeks since prior cytokines
* More than 4 weeks since prior plasmapheresis or plasma exchange
* No prior stem cell or bone marrow transplant

Chemotherapy:

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas, mitomycin, or high-dose carboplatin)
* No prior intensive chemotherapy with stem cell support

Endocrine therapy:

* More than 4 weeks since prior corticosteroids
* No concurrent corticosteroids

Radiotherapy:

* More than 4 weeks since prior radiotherapy involving more than 25% of bone marrow

Surgery:

* Recovered from any prior surgery
* No prior organ transplant

Other:

* No other concurrent investigational agent
* No concurrent immunosuppressants
* No concurrent anti-inflammatory agents including aspirin and non-steroidal anti-inflammatory agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-03

CONTACTS AND LOCATIONS:
Overall Officials: Suzin Mayerson, PhD, Study Chair — LifeTime Pharmaceuticals
Locations (1):
- Victory Over Cancer, Rockville, Maryland, United States